CLINICAL TRIAL: NCT01427374
Title: Clinical, Biochemical and Genetic Risk Factors for Coronary Artery Calcification and Left Ventricular Hypertrophy in Hemodialysis Patients (CKDCS/LUCID)
Brief Title: Risk Factors for Coronary Artery Calcification and Left Ventricular Hypertrophy in Hemodialysis Patients
Status: Terminated | Type: Observational
Why Stopped: low recruitment
Sponsor: University of Alberta (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marcello Tonelli, MD, Associate Professor, University of Alberta
Other Study IDs: 2011P000387; IRO 90262 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; peritoneal dialysis; chronic kidney disease; cardiovascular risk factors; cardiac imaging; dialysis; parathyroid hormone; vitamin D; coronary artery calcification; left ventricular hypertrophy; genetic predisposition; biochemical markers; infection; pharmacogenomics
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular; Genetic Predisposition to Disease; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine will be obtained at baseline, 6 months and annually thereafter. Blood samples will be immediately divided into multiple aliquots, from which plasma, DNA, RNA and/or cells will be extracted and separately stored. Urine specimens will also be aliquoted to allow future measurement of genetic and cellular material. Specimens will be labeled using unique study identifiers to maintain confidentiality.
Oversight: Data Monitoring Committee: No

SUMMARY:
Individuals with kidney disease are at a higher risk for heart and vascular diseases, including heart attacks and strokes, than those with normal kidney function. The purpose of this research study is to collect information on the causes, complications and treatment of kidney disease. Patient characteristics, comorbid diseases and laboratory markers used in routine practice, as well as novel biochemical markers and genetic data will be collected to examine relationships between biochemical and genetic markers and cardiovascular risk. Information on the health history of incident hemodialysis and peritoneal dialysis patients will be captured using structured patient interviews and review of medical records. Blood and urine specimens will be collected at the time of dialysis initiation and stored in order to perform novel biochemical and genetic assays in the future. The overall goal of the CKDCS/LUCID study is improve understanding of cardiac-associated risks and to improve treatment in patients with kidney disease. A cardiac imaging substudy will be performed in a subset of patients enrolled. The goals of the substudy are to examine whether the risks of developing common cardiac-related complications (coronary artery calcification [CAC] and left ventricular hypertrophy [LVH]) are associated with certain medications taken by individuals on dialysis and whether these risks are modified by a genotypic predisposition.

DETAILED DESCRIPTION:
This study is being conducted under the Sponsorship of the University of Alberta (Edmonton, Alberta, Canada) and is funded by Canadian Institutes of Health Industry Partnered Research Grant IRO 90262 - with partnership funding from Abbott Laboratories. The co-Principal Investigators are Marcello Tonelli MD SM and Ravi Thadhani, MD, MPH . A total of 750 patients are anticipated being enrolled at Massachusetts General Hospital (MGH). The remaining patients are being enrolled in Canada.

This study will utilize data from "The Canadian Kidney Disease Cohort Study" (CKDCS) and "The Longitudinal US/Canada Incident Dialysis STUDY (LUCID).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age) commencing hemodialysis or peritoneal dialysis.

Exclusion Criteria:

• Unable to provide informed consent.

Exclusion Criteria for the cardiac substudy:

CT exclusion criteria

1. Pregnancy
2. Obesity (>275 lbs)
3. Rapid atrial fibrillation, bigeminy or trigeminy
4. Any condition that impedes the ability to lie flat during the CT (eg:decompensated congestive heart failure).

MRI exclusion criteria

1. Cardiac pacemaker or implantable defibrillator
2. Obesity (>275lbs)
3. Intraocular metal
4. Cerebral aneurysm clips, programmable shunt, etc.
5. Any type of ear implant
6. Any implanted device (eg: insulin, drug infusion device)
7. Metal shrapnel or bullet
8. Any condition that impedes the ability to lie flat during the MRI (eg:decompensated congestive heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident hemodialysis and peritoneal dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Calcification | baseline

SECONDARY OUTCOMES:
Coronary Artery Calcification | 12 months
Left ventricular mass | baseline
Left ventricular mass | 12 months
All cause mortality | 12 months
Left ventricular hypertrophy | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital; Marcello Tonelli, MD, SM, FRCP, Principal Investigator — University of Alberta
Locations (4):
- United States (3):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Washington, Seattle, Washington
- University of Alberta, Edmonton, Alberta, Canada